CLINICAL TRIAL: NCT06895616
Title: Effect of Baseline Cortisol Level on Lipid Peroxidation Products in Young Female Swimmers
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: SWIMMER- 2024
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Stress Oxidative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Eppendorf tubes with serum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Research group: twenty-four and homogeneous female swimmers, who train swimming intensively and attend the Sports Championship School Complex. In this cohort, baseline serum cortisol levels were considered, and the athletes were divided into two groups: 1) Serum cortisol <230 (normal): n=14 2) Serum cortisol >230 ng/ml (high): n=10

In this study, the athletes were subjected to intensive swimming tests in breaststroke crawl (800m + 200m + 50m) with 15 minutes of active rest between test sections in the water.

Blood samples took from the cubital vein at three time points: before stress test (pre-exercise), one minute after the end of the test (post-exercise), and after a 3-hour recovery period (3h recovery). Measurements morphology, 4-Hydroxynonenal (4-HNE), 8-isoprostane, cortysol levels were determined using ELISA kits.

DETAILED DESCRIPTION:
The data of 24 trained female from the Sports Championship School Complex. All athletes presented as medically fit, with no underlying health problems. In this cohort, baseline serum cortisol levels were considered, and the athletes were divided into two groups: 1) Serum cortisol <230 (normal): n=14 2) Serum cortisol >230 ng/ml (high): n=10 In this study, the athletes were subjected to intensive swimming tests in breaststroke crawl (800m + 200m + 50m) with 15 minutes of active rest in the water. Blood samples took from the cubital vein at three time points: before stress test (pre-exercise), one minute after the end of the test (post-exercise), and after a 1-hour recovery period (3h recovery).

Measurement: All determined parameters were measured with the available equipment in the ZWKF laboratory in Gorzów Wielkopolski and using commercial assay kits. Measurements were performed by the project contractors.

1. Polyethylene tubes (2.7ml) containing dipotassium ethylenediaminetetraacetic acid (EDTAK2) anticoagulant were used for the following tests: (a) complete blood count (7 parameters) determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland). Red blood cell indices: RBC (Red Blood Cells), HGB (Hemoglobin), HCT (Hematocrit), MCV (Mean Corpuscular Volume), MCH (Mean Corpuscular Hemoglobin), MCHC (Mean Corpuscular Hemoglobin Concentration), RDW (Red Blood cells Distribution Width). (b) a manual blood smear was made by placing a drop of blood on a slide and then spreading it with a uniform motion. After drying, it was colored by the May Grunwald-Giemsa method according to the procedure. The stained and fixed smear after drying was viewed under a microscope for quantitative and qualitative assessment.
2. Polyethylene clotting activator tubes (9 ml) were centrifuged to separate the morphotic elements from the serum using a centrifuge (3000 rpm for 10 min). The serum was pipetted into several Eppendorf tubes, which then was frozen (temp. -80 °C). All the following biochemical parameters were determined from the extracted serum: (a) using the ELISA method by the test manufacturer's instructions. The designations include the flowing parameters:

4-Hydroxynonenal (4-HNE), 8-isoprostane, cortysol. (3) The lactate (La) concentration was determined from the capillary blood immediately after collection using a commercially available kit (Dr. Lange, Germany).

The athletes' diets were completely analyzed before each exercise test by a nutritionist. Participants, with the help of a dietician who was available during meals on test days, filled out food diaries. The amount of energy, protein, carbohydrates, fats and fiber were then analyzed using a commercially available program.

The experiment was conducted in accordance with the Declaration of Helsinki. The study protocol was approved by the Ethical Committee of the Medical University of Poznan

ELIGIBILITY:
Inclusion Criteria:

* valid medical examination,
* consent of the legal guardian of the underage athlete to participate in the study,
* Training experience a minimum of three years
* Student of a sports championship school team,
* ompletion of the exercise test in the swimming pool - crawl style intensive test (800 m + 200 m + 50 m) on two test deadline

Exclusion Criteria:

* antibiotic therapy,
* supplementation, use of any drugs or oral hormonal contraceptives
* health problems within the last months

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Swimmers attending the Sports Championship School Complex
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in 4-Hydroxynonenal (4-HNE) level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of 4-Hydroxynonenal (4-HNE) [pg/ml]. ELISA method by the test manufacturer's instructions
Changes from baseline in 8-isoprostane level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of 8-isoprostane [ng/mL]. ELISA method by the test manufacturer's instructions
Changes from baseline in Cortysol level. | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  Concentration of cortysol [ng/mL]. ELISA method by the test manufacturer's instructions
a manual blood smear | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  was made by placing a drop of blood on a slide and then spreading it with a uniform motion. After drying, it was colored by the May Grunwald-Giemsa method according to the procedure. The stained and fixed smear after drying was viewed under a microscope for quantitative and qualitative assessment.
complete blood count | At rest (before the test), directly after the test, and after a 3-hour recovery period.
  erythrocytes: RBC [10^6/mL], HGB [g/dL], HCT [%], MCV [mm^3], MCH [pg], MCHC [g/dL], RDW [%].

SECONDARY OUTCOMES:
Antropometric characteristic - height | Day 1 after overall fast
  Prior to the exercise test, the investigator measured the anthropometric parameters, including height (Seca 213 Hamburg, Deutschland) [cm]
Antropometric characteristic - weight | Day 1 after overall fast
  Prior to the exercise test, the investigator measured the anthropometric parameters, including weight (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [kg]
Food record - energy | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program: energy [kcal]
Food record - protein | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program: protein [kcal]
Food record - carobhydrates | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record.The results were calculated using the dietetykpro program: carobhydrates [kcal]
Food record - fiber | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program: fiber [kcal]
Food record - fat | Day before the Day 1, in the morning at Day 1
  Participants prepared a food record. The results were calculated using the dietetykpro program: fat [kcal]

CONTACTS AND LOCATIONS:
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No